CLINICAL TRIAL: NCT06670963
Title: The Use of Epoetin Alfa and Iron Derisomaltose in the Treatment of Anemia in Patients With Sepsis or Septic Shock Hospitalized in the Intensive Care Unit: a Randomized Controlled Clinical Trial
Brief Title: Use of Epoetin Alfa and Iron Derisomaltose in Treatment of Anemia in Patients With Sepsis or Septic Shock: a Randomized Controlled Trial
Acronym: EpoAid
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Piotr Czempik (Other)
Responsible Party: Sponsor-Investigator, Piotr Czempik, Assistant Professor, MD, PhD, Medical University of Silesia
Organization: Medical University of Silesia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BNW-1-006/N/4/K
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Anemia; Sepsis; Septic Shock
Keywords: anemia; sepsis; septic shock; epoetin alfa; iron derisomaltose; red blood cell; hemoglobin; intensive care unit
MeSH Terms: conditions — Anemia; Sepsis; Shock, Septic | interventions — Iron; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epoetin alfa +/- ferric derisomaltose (Experimental): Epoetin alfa 50 units/kg IV 3 times weekly and ferric derisomaltose 0.2g IV if reticulocyte hemoglobin equivalent <29.3 pg
  Interventions: Drug: Iron; Drug: EPO
- Placebo (Placebo Comparator): 0.9% NaCl
  Interventions: Drug: 0.9 % NaCl

INTERVENTIONS:
Drug: Iron — Iron derisomaltose 0.2g IV if reticulocyte hemoglobin equivalent <29.3 pg (lower limit for the local laboratory reference range for reticulocyte hemoglobin equivalent)
  Arms: Epoetin alfa +/- ferric derisomaltose
Drug: EPO — Epoetin alfa 50 units/kg IV 3 times weekly
  Arms: Epoetin alfa +/- ferric derisomaltose
Drug: 0.9 % NaCl — Volume of 0.9% NaCl identical as volume of medications used in experimental arm
  Arms: Placebo

SUMMARY:
Background Up to 66% of have anemia at the admission to the intensive care unit. This number increases to 95% after 72 hours of hospitalization in the intensive care unit due to illness and iatrogenic blood loss. Anemia worsens tissue oxygenation, especially in patietns with sepsis or septic shock, who already have blood flow issues. Instead of giving blood transfusions, which can have side effects, we aim to address the root causes of anemia in these patients. Sepsis can cause "inflammatory anemia" and combine with iron deficiency anemia. Current anemia treatments include drugs that stimulate red blood cell production and intravenous iron supplements. Some think that iron supplements can worsen infections by feeding pathogens, but this is not conclusively proven. Since transfused red blood cells (RBC) also contain iron, small doses of intravenous iron might help sepsis patients with iron deficiency.

There is a need for a study on the effects of epoetin alfa and iron derisomaltose on hemoglobin (Hb) levels in sepsis patients.

Hypothesis and Aim Treating anemia in sepsis patients could increase Hb levels and reduce RBC transfusions, improving patient outcomes. This study aims to evaluate the effects of epoetin alfa ± iron derisomaltose on Hb levels and RBC transfusion rates.

Primary Endpoints:

1. Hb difference at study exit (discharge from ICU/death/bleeding/need for surgery/day 15 whatever comes first) and day 1 corrected for Hb increase due to possible RBC transfusion

Secondary Endpoints:

1. Hb difference on days 8 and 1 corrected for Hb increase due to possible RBC transfusion
2. Hb difference on days 15 and 1 corrected for Hb increase due to possible RBC transfusion
3. number of blood transfusions
4. percentage of patients receiving at least one blood transfusion
5. actual vs. predicted mortality
6. prevalence of deep vein thrombosis and pulmonary embolism
7. mortality rates in ICU, hospital, 30-day, and 90-day.

Materials and Methods:

This will be a randomized controlled clinical trial recruting 200 patients

Inclusion Criteria:

1. age ≥18
2. diagnosed sepsis (Sepsis-3 definition) or septic shock (Septic Shock-3 definition)
3. hemoglobin <120 g/L for both sexes

Exclusion Criteria:

1. bleeding
2. decompensated liver disease
3. inherited microcytic disorders
4. macrocytosis
5. contraindications to pharmacological prophylaxis for venous thromboembolism
6. pregnancy
7. allergy to epoetin alfa and/or iron derisomaltose.
8. ferritin >800 ng/mL.
9. inability to take consent

Study Group:

1. epoetin alfa 50 u/kg IV (days 1, 3, 5, 8, 10, 12)
2. iron derisomaltose 0.2g IV when RET-He <29.3 pg (days 1, 3, 5, 8, 10, 12)
3. algorithm for red blood cell transfusions

Control Group:

1. algorithm for red blood cell transfusions

Laboratory Parameters:

Initial: interleukin-6, procalcitonin, C-reactive protein, creatinine, ammonia, blood urea nitrogen, aspartate aminotransferase, alanine aminotransferase, total bilirubin, complete blood count (CBC), reticulocytes (RET), ferritin, iron, transferrin.

Serial: CBC and RET (days 1, 3, 5, 8, 10, 12)

DETAILED DESCRIPTION:
Project Description:

Project Title: The use of epoetin alfa and iron derisomaltose in treating anemia in patients with sepsis or septic shock in the ICU: a randomized controlled clinical trial.

Project Acronym: EpoAid

Theoretical Background and Rationale: Up to 66% of patients have anemia at admission to the intensive care unit. Additionally, many patients develop anemia during hospitalization in the intensive care unit due to illness and iatrogenic blood loss for laboratory diagnostics. After 72 hours 95% of intensive care unit patients are anemic. Anemia increases the risk of tissue oxygen deficiency, which is particularly important in sepsis or septic shock patients who may have peripheral perfusion disorders due to infection. Anemia should be treated causally because red blood cell transfusions can lead to adverse effects, including immunomodulation leading to innate immunity suppression, which is particularly significant in critically ill sepsis or septic shock patients. Anemia caused by sepsis is known as inflammatory anemia (AI). Sepsis patients often have mixed anemia, combining features of AI and iron deficiency anemia (IDA) - AI+IDA. Currently available treatments for mixed anemia include erythropoiesis-stimulating agents (ESA) and intravenous iron supplements (e.g., iron derisomaltose). Manufacturers of intravenous iron products contraindicate their use in infections since intravenous iron could theoretically exacerbate infections by stimulating pathogen growth. However, there is no conclusive data on this. Considering that stored red blood cells are also a source of iron that pathogens can use, it seems that fractional doses of intravenous iron could benefit sepsis patients with diagnosed iron deficiency. Additionally, ESA administration could cause functional iron deficiency, where small doses of intravenous iron might also be beneficial.

Attempts to use ESA and intravenous iron in the general ICU population have yielded inconclusive results due to methodological errors. In the IRONMAN study comparing iron carboxymaltose with placebo, no difference in transfusion rates (primary endpoint) was found, but higher Hb levels were observed at hospital discharge in the intervention group (107 vs. 100 g/L). This trial had some methodological flaws: intravenous iron was administered regardless of anemia etiology, red blood cell transfusion decisions were made by clinicians - there was no transfusion algorithm, and the average hospital stay was 11 days - maximal effect of intravenous iron is seen after 3-4 weeks, at least 2 weeks.

Iron deficiency diagnostics in sepsis patients must rely on parameters independent of the systemic inflammatory response since standard iron metabolism parameters (ferritin, transferrin saturation) are not useful here. Severe sepsis was an exclusion criterion in the IRONMAN study. Given the limitations of previous studies and the lack of research on the use of intravenous iron in sepsis patients, it is warranted to conduct a study evaluating the effect of epoetin alfa ± iron derisomaltose on Hb levels in sepsis or septic shock patients.

Hypothesis and Research Aim: Causal treatment of anemia in sepsis or septic shock patients may lead to increased Hb levels and reduced transfusion rates, potentially improving patient outcomes. This study aims to evaluate the effect of epoetin alfa ± iron derisomaltose on one primary and several secondary outcomes.

Materials and Methods: A randomized controlled clinical trial is planned. Blinding will be single due to the color (rusty) of the intervention drug (iron derisomaltose) and problems with complete blinding of the intervention. Randomization will be done using a computer generator of randomized numbers using block of 4. Two hundred patients will be recruited (100 in the experimental group, 100 in the control group). If a study subject starts bleeding or requires surgery (affects Hb levels and transfusion necessity - primary endpoints), the time until this event will be evaluated. Data collected: demographics (gender, age), infection site, length of stay (ICU, hospital), mortality (ICU, hospital, 30 days, 90 days). Blood loss for laboratory diagnostics will be monitored (calculation based on laboratory parameters ordered and test tube used). Pharmacological venous thromboembolism prophylaxis will be used in the experimental and contorol groups: enoxaparin 40 mg x 1 sc in patients with creatinine clearance ≥30 mL/min or dalteparin 5000 IU x 1 sc in patients with creatinine clearance <30 mL/min, and a red blood cell transfusion decision algorithm will be employed.

Experimental group:

1. epoetin alfa (Binocrit, Sandoz, Poland) given intravenously when Hb <120 g/L, dosed by a study subject weight:

   * 2000 IU (<60 kg)
   * 3000 IU (60-79 kg)
   * 4000 IU (80-99 kg)
   * 5000 IU (>100 kg) administered on days 1, 3, 5, 8, 10, 12
2. iron derisomaltose (Monover, Pharmacosmos, Denmark) given intravenously at a dose of 0.2g when Hb <120 g/L and RET-He <29.3 pg, administered on days 1, 3, 5, 8, 10, 12
3. red blood cell transfusion decision based on a proprietary decision algorithm. Binocrit will be stored at 2-8 °C. Before use, the drug will be stored at room temperature for 15 minutes. The drug is packaged in prefilled syringes; it will be mixed with 0.9% sodium chloride to a volume of 20 mL, then injected intravenously as a bolus, followed by a 20 mL 0.9% NaCl sodium chloride bolus to ensure immediate drug entry into the bloodstream. It is crucial to administer the entire dose without loss, as it is the primary intervention drug in this study. Monover is provided in 0.1g ampoules. The drug will be administered at a fixed dose of 0.2g when RET-HE <29.3 pg on the scheduled administration day. The drug will be diluted with 0.9% NaCl to a volume of 50mL and administered in a brown 50mL syringe using an infusion pump at a rate of 60mL/h.

Control Group:

red blood cell transfusion decision based on a proprietary decision algorithm.

Monitored parameters:

* initial lab parameters (extended): interleukin-6, procalcitonin, C-reactive protein, creatinine, ammonia, blood urea nitrogen, aspartate aminotransferase (AspAT), alanine aminotransferase, total bilirubin, complete blood count (CBC), reticulocytes (RET), ferritin, iron, transferrin.
* serial measurements: Hb and hemoglobin equivalent in reticulocytes (RET-He) on the day of epoetin alfa ± iron derisomaltose administration.

Timeline: November 2024 - December 2026

Feasibility: given the number of ICU hospitalizations (approximately 400 per year) and the prevalence of sepsis/septic shock, it will be possible to enroll about 100 patients per year.

ELIGIBILITY:
Inclusion criteria:

1. age ≥18,
2. diagnosed sepsis (Sepsis-3) or septic shock (Septic Shock-3),
3. hemoglobin <120 g/L in both sexes.

Exclusion criteria:

1. bleeding,
2. decompensated liver disease,
3. inherited microcytic disorders,
4. macrocytosis,
5. contraindications to pharmacological prophylaxis of VTE,
6. pregnancy,
7. allergy to epoetin alfa and/or iron derisomaltose,
8. ferritin concentration >800 ng/mL,
9. unable to take informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin concentration difference at exit from the study | From enrollment to day 15/death/discharge from ICU/bleeding episode/surgery whatever comes first
  The difference between hemoglobin concentration at exit from the study and day 1 corrected for Hb increase due to possible RBC transfusion [RBC volume x RBC Hb concentration/study subject's blood volume (weight x 65 mL for women/weight x 75 mL for men)]

SECONDARY OUTCOMES:
Hemoglobin concentration difference at 1 week | From enrollment to day 8 (if a study subject still in the trial)
  The difference in hemoglobin concentration on days 8 and 1 corrected for Hb increase due to possible RBC transfusion [RBC volume x RBC Hb concentration/study subject's blood volume (weight x 65 mL for women/weight x 75 mL for men)]
Hemoglobin concentration difference at 2 weeks | From enrollment to day 15 (if a study subject still in the trial)
  The difference in hemoglobin concentration between day 15 and day 1 corrected for Hb increase due to possible RBC transfusion [RBC volume x RBC Hb concentration/study subject's blood volume (weight x 65 mL for women/weight x 75 mL for men)]
Number of red blood cell units transfused | From enrollment to day 15/death/discharge from ICU/bleeding episode/surgery whatever comes first
  Number of allogeneic red blood cell units transfused
Tranfusion rate | From enrollment to day 15/death/discharge from ICU/bleeding episode/surgery whatever comes first
  Percentage of study subjects receiving at least one red blood cell unit
Deep vein thrombosis prevalence | From enrollment to day 15/death/discharge from ICU/bleeding episode/surgery whatever comes first
  Number of deep vein thrombosis cases
Pulmonaly embolism prevalence | From enrollment to day 15/death/discharge from ICU/bleeding episode/surgery whatever comes first
  Number of pulmonary embolism cases
Intensive care unit mortality | From enrollment to discharge from ICU
  Death during intensive care unit hospitalization (index hospitalization)
30-day mortality | From enrollment to day 30
  Death within 30 days of day 1
90-day mortality | From enrollment to day 90
  Death within 90 days of day 1
Actual vs. predicted intensive care unit mortality | From enrollment to discharge from ICU
  Difference between actual intensive care unit mortality and intensive care unit mortality predicted by Sequential Organ Failure Assessment Score (index hospitalization)
Actual vs. predicted intensive care unit mortality | From enrollment to discharge from ICU
  Difference between actual intensive care unit mortality and intensive care unit mortality predicted by Acute Physiology And Chronic Health Evaluation Score (index hospitalization)
Actual vs. predicted intensive care unit mortality | From enrollment to discharge from ICU
  Difference between actual intensive care unit mortality and intensive care unit mortality predicted by Simplified Acute Physiology Score III (index hospitalization)

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersyteckie Centrum Kliniczne im. prof. K. Gibińskiego Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No
Data privacy issues

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] IRONMAN Investigators; Litton E, Baker S, Erber WN, Farmer S, Ferrier J, French C, Gummer J, Hawkins D, Higgins A, Hofmann A, De Keulenaer B, McMorrow J, Olynyk JK, Richards T, Towler S, Trengove R, Webb S; Australian and New Zealand Intensive Care Society Clinical Trials Group. Intravenous iron or placebo for anaemia in intensive care: the IRONMAN multicentre randomized blinded trial : A randomized trial of IV iron in critical illness. Intensive Care Med. 2016 Nov;42(11):1715-1722. doi: 10.1007/s00134-016-4465-6. Epub 2016 Sep 30. PMID 27686346
- [Background] Czempik PF, Wilczek D, Herzyk J, Krzych LJ. Hospital-Acquired Anemia in Patients Hospitalized in the Intensive Care Unit: A Retrospective Cohort Study. J Clin Med. 2022 Jul 6;11(14):3939. doi: 10.3390/jcm11143939. PMID 35887702
- [Background] Czempik PF, Pluta MP, Krzych LJ. Physiologic approach to red blood cell transfusion in non-bleeding critically ill patients. Arch Med Sci. 2022 Aug 30;18(5):1423-1425. doi: 10.5114/aoms/152217. eCollection 2022. No abstract available. PMID 36160360
- [Background] Czempik PF, Wiorek A. Comparison of Standard and New Iron Status Biomarkers: A Prospective Cohort Study in Sepsis Patients. Healthcare (Basel). 2023 Mar 30;11(7):995. doi: 10.3390/healthcare11070995. PMID 37046922
- [Background] Czempik PF, Wiorek A. Iron deficiency in sepsis patients managed with divided doses of iron dextran: a prospective cohort study. Sci Rep. 2023 Mar 31;13(1):5264. doi: 10.1038/s41598-023-32002-y. PMID 37002279
- [Background] Czempik PF, Wiorek A. Iron deficiency in sepsis patients based on reticulocyte hemoglobin and hepcidin concentration: a prospective cohort study. Arch Med Sci. 2023 May 24;19(3):805-809. doi: 10.5114/aoms/161802. eCollection 2023. PMID 37313179